CLINICAL TRIAL: NCT02159326
Title: Microgynon Riociguat Drug Interaction Study to Investigate the Effect of Riociguat 2.5 mg 3 Times Daily Multiple-dose Treatment on the Plasma Concentrations of / Exposure to Levonorgestrel and Ethinyl Estradiol in Healthy Postmenopausal Women in a 2-fold Crossover Design
Brief Title: Microgynon Riociguat Drug Interaction Study in Healthy Postmenopausal Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 17309; 2014-000829-20 (EudraCT Number)
Record Dates: First submitted 2014-06-06; First posted 2014-06-09 (Estimated); Last update posted 2015-08-14 (Estimated); Status verified 2015-08

CONDITIONS: Drug Interactions
MeSH Terms: interventions — ethinyl estradiol, levonorgestrel drug combination; riociguat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm1 (Experimental): single oral tablet dose of Microgynon (0.03 mg EE and 0.15 mg LNG, fasted)
  Interventions: Drug: Microgynon
- Arm2 (Experimental): multiple oral tablet doses of 2.5 mg riociguat TID over 12 days and, on the seventh day of this treatment, a single oral tablet dose of Microgynon (0.03 mg EE and 0.15 mg LNG, fasted)
  Interventions: Drug: Microgynon; Drug: Riociguat (Adempas,BAY63-2521)

INTERVENTIONS:
Drug: Microgynon — single oral tablet dose of Microgynon (0.03 mg EE and 0.15 mg LNG, fasted)
Drug: Riociguat (Adempas,BAY63-2521) — multiple oral tablet doses of 2.5 mg riociguat TID over 12 days and, on the seventh day of this treatment
  Arms: Arm2

SUMMARY:
Physicians might be concerned that Adempas may have a metabolic interaction with oral contraceptives (OC) that could decrease the contraceptive efficacy of the OC. The information regarding lack of potential pharmacokinetic interaction has been communicated; there is a need for more re-assurance and further data that there is no interaction between Adempas and OCs. A drug-drug interaction study of riociguat with an OC such as Microgynon in the least vulnerable population for these purposes, i.e. healthy postmenopausal women, is considered adequate to inform about safe use of Adempas with OCs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subject
* Non-smokers of at least 3 month before screening
* Age: 52 to 65 years (inclusive) at the first screening examination
* Ethnicity: white
* Body mass index (BMI)>=20 and <=32 kg/m2
* Postmenopausal state, defined as
* Medical history, if applicable (natural menopause at least 12 months before the first study drug administration and hormone analyses in serum
* Age<60 years: follicle-stimulating hormone (FSH) >40 IU/L in plasma
* Age <60 years: estradiol (E2) <20 ng/L (<73 pmol/L) in plasma

Exclusion Criteria:

* History of coronary artery disease, Symptomatic postural hypotension, History of bronchial asthma, known hypersensitivity to the study, relevant diseases within 4 weeks before study drug administration,
* Presence or a history of venous or arterial thrombotic / thromboembolic events or cerebrovascular accident, a high risk for venous or arterial thrombosis,
* Use of systemic or topical medicines or substances which oppose the study objectives, smoking, use of sex hormones in any forms
* Clinically relevant findings in the ECG, systolic blood pressure below 110 or above 145 mmHg, heart rate below 50 or above 95 beats per minute
* Clinically relevant findings in the gynecological examination,
* Participation in another clinical study

Ages: 52 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-06; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time curve (AUC) of Ethinylestradiol (EE) | Up to 4 months
  Plasma concentrations Ethinyl estradiol (EE) and levonorgestrel (LNG)
Area under the plasma concentration time curve (AUC) of Levonorgestrel (LNG) | Up to 4 months
Maximal concentration (Cmax) of Ethinylestradiol (EE) | Up to 4 months
Maximal concentration (Cmax) of Levonorgestrel (LNG) | Up to 4 months

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | Up to 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Mönchengladbach, North Rhine-Westphalia, Germany